CLINICAL TRIAL: NCT06468592
Title: Implantation in the Palatal Process of the Maxilla as a Modification of the Osteotome Sinus Floor Elevation (Summers Technique)
Brief Title: Implantation in Posterior Maxilla in Cases With Insufficient Bone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UDDS-OMFS-1-2024
Record Dates: First submitted 2024-06-15; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Bone Loss in Jaw; Implant Site Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tilted implants (Experimental): The tilted implants are inserted palatally into the maxillary sinus
  Interventions: Procedure: Tilted insertion of implants
- Straight implants (Active Comparator): The implants inserted into the maxillary sinus in an axial direction
  Interventions: Procedure: Straight insertion of implants

INTERVENTIONS:
Procedure: Tilted insertion of implants — Using osteotomes, implants are inserted and tilted from 30° to 45° into the palatal direction from the maxillary sinus.
  Arms: Tilted implants
Procedure: Straight insertion of implants — The implants are inserted in an axial direction into the maxillary sinus according to Summers' traditional technique.
  Arms: Straight implants

SUMMARY:
Dental implant procedures are performed on two groups of individuals who share the common characteristic of insufficient bone for traditional implantation.

The first group lacks a palatal process, while the second group has a palatal process. Then, compare the initial primary stability of implants in the maxillary bone-type (D4) that were inserted tilted in the palatal process of the maxilla, palatally from the maxillary sinus, with implants inserted axially into the maxillary sinus by using a manual torque wrench.

DETAILED DESCRIPTION:
Increasing the initial primary stability intensity value increases the success rate of implants in general and also allows immediate or early loading procedures to begin. In addition, to avoid complications resulting from inserting implants into the compromised maxillary sinus according to the Summers method. The most important of these is perforation of the mucous membrane lining the maxillary sinus and the possibility of its application in pathological cases of the maxillary sinus, such as chronic maxillary sinusitis and the presence of mucous retention cysts, in which intervention according to the usual Summers method is not indicated.

Despite the previous advantages obtained by this method, there are some disadvantages to the technique of tilting the implants in the palatal direction from the maxillary sinus, which are the limitation of its application to cases with a palatal process of the maxilla in the upper jawbone, which requires performing a three-dimensional radiograph. It was observed in this study and after studying the cross-sections that sufficient thickness for this process was less likely present than in cases of its absence. In addition, prosthetic procedures are generally difficult in tilted implants compared to axial implants.

ELIGIBILITY:
Inclusion criteria for both groups:

* Patients must have inadequate bone density in the posterior region of the upper jaw.
* Patients should maintain good oral hygiene.
* The surgical site must be free from infection.
* There should be no contraindications for oral surgery.

For the first group:

- Patients in the first group must have a palatal process of the maxillary bone determined by radiographic examination.

Exclusion criteria:

* Patients with adequate bone volume to receive an implant.
* Patients with systemic diseases that impair metabolism or healing at the surgical site.
* Patients with contraindications for surgery, including cardiovascular disorders, blood clotting disorders, anticoagulant use, or uncontrolled diabetes.
* Patients receiving medications that affect bone metabolism, such as corticosteroids, oral contraceptives, hormonal treatments, or those undergoing chemical or radiological therapies.

Ages: 32 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
The initial implant stability | one time assessment at five minutes following the completion of inserting implants.
  Primary stability was recorded for all implants in both groups, estimated by Newton/cm (N/cm), using a manual torque wrench.
  This manual measure consists of a fixed arm installed above the implants and a moving arm moving away from the fixed arm in a clockwise direction, graduating from 5-45 Newtons. When the moving arm stops, the distance between it and the fixed arm expresses the first degree of the initial primary stability.

CONTACTS AND LOCATIONS:
Locations (1):
- Orthodontics Department, Faculty of Dentistry, University of Aleppo, Aleppo, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Summers RB. The osteotome technique: Part 2--The ridge expansion osteotomy (REO) procedure. Compendium. 1994 Apr;15(4):422, 424, 426, passim; quiz 436. PMID 8055514
- [Background] Summers RB. The osteotome technique: Part 3--Less invasive methods of elevating the sinus floor. Compendium. 1994 Jun;15(6):698, 700, 702-4 passim; quiz 710. PMID 7994726
- [Background] Summers RB. The osteotome technique: Part 4--Future site development. Compend Contin Educ Dent. 1995 Nov;16(11):1090, 1092 passim; 1094-1096, 1098, quiz 1099. PMID 8598008
- [Background] Boyne PJ. Analysis of performance of root-form endosseous implants placed in the maxillary sinus. J Long Term Eff Med Implants. 1993;3(2):143-59. PMID 10146541
- [Background] Del Fabbro M, Ceresoli V. The fate of marginal bone around axial vs. tilted implants: a systematic review. Eur J Oral Implantol. 2014 Summer;7 Suppl 2:S171-89. PMID 24977252
- [Background] Barnea E, Tal H, Nissan J, Tarrasch R, Peleg M, Kolerman R. The Use of Tilted Implant for Posterior Atrophic Maxilla. Clin Implant Dent Relat Res. 2016 Aug;18(4):788-800. doi: 10.1111/cid.12342. Epub 2015 Apr 8. PMID 25853626
- [Background] Malo P, de Araujo Nobre M. Partial rehabilitation of the posterior edentulous maxilla using axial and tilted implants in immediate function to avoid bone grafting. Compend Contin Educ Dent. 2011 Nov-Dec;32(9):E136-45. PMID 23627307
- [Background] Penarrocha-Oltra D, Candel-Marti E, Ata-Ali J, Penarrocha-Diago M. Rehabilitation of the atrophic maxilla with tilted implants: review of the literature. J Oral Implantol. 2013 Oct;39(5):625-32. doi: 10.1563/AAID-JOI-D-11-00068. Epub 2011 Nov 28. PMID 22121829
- [Background] Bruschi E, Manicone PF, De Angelis P, Papetti L, Pastorino R, D'Addona A. Comparison of Marginal Bone Loss Around Axial and Tilted Implants: A Retrospective CBCT Analysis of Up to 24 Months. Int J Periodontics Restorative Dent. 2019 Sep/Oct;39(5):675-684. doi: 10.11607/prd.4110. PMID 31449578